CLINICAL TRIAL: NCT00514020
Title: Pharmacogenomically Selected Treatment for Gastric and Gastroesophageal Junction (GEJ) Tumors: A Phase II Study
Brief Title: Fluorouracil, Oxaliplatin, and Leucovorin in Treating Patients With Metastatic Stomach Cancer or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Laura W. Goff, MD, Assistant Professor of Medicine; Associate Director, Hematology/Oncology Fellowship Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 0716; P30CA068485 (NIH); VU-VICC-GI-0716
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Results first posted 2012-10-18 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Gastric Cancer
Keywords: adenocarcinoma of the stomach; stage IV gastric cancer; recurrent gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Genetic: gene expression analysis; Genetic: polymorphism analysis; Genetic: protein expression analysis; Other: pharmacological study

INTERVENTIONS:
Drug: fluorouracil — Given through a vein over 5 minutes and then continuously over 46 hours on days 1 and 15.
Drug: leucovorin calcium — through a vein over 2 hours on days 1 and 15.
Drug: oxaliplatin — 500 ml D5W through a vein over 2 hours on days 1 and 15.
Genetic: gene expression analysis — Blood collection
Genetic: polymorphism analysis — Blood collection
Genetic: protein expression analysis — Blood collection
Other: pharmacological study — Blood collection

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, oxaliplatin, and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving fluorouracil together with oxaliplatin and leucovorin works in treating patients with metastatic stomach cancer or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the response rate in patients with "good risk" genotype (TSER*2/*2 or TSER*2/*3 genotype [low TS expression]) to historical control response rates in non-genotype selected patients.

OUTLINE: This is a multicenter study.

Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 5 minutes and then continuously over 46 hours on days 1 and 15. Courses repeat every 2 weeks in the absence of unacceptable toxicity or disease progression.

Available tumor tissue samples are assessed for expression of TS at the mRNA and protein levels. The results are correlated with germline and tumor TSER genotypes as well as response to the study treatment regimen. Polymorphisms in other genes associated with treatment outcome or toxicity are also assessed.

After completion of study treatment, patients are followed periodically for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal junction

  * Metastatic disease
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan
* No known active brain metastases

  * Patients with treated brain metastases are eligible if stable off steroids for at least 30 days

PATIENT CHARACTERISTICS:

* ECOG performance status ≤ 2 (Karnofsky performance status ≥ 60%)
* Life expectancy ≥ 3 months
* WBC ≥ 3,000/μL
* Absolute neutrophil count ≥ 1,500/μL
* Platelets ≥ 100,000/μL
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* AST or ALT ≤ 2.5 x ULN (< 5 x ULN if known liver metastases)
* Creatinine clearance ≤ 1.5 x ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 21 days after completion of study treatment
* No history of allergic reactions to fluorouracil or oxaliplatin
* No concurrent uncontrolled illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* No prior therapy for metastatic disease

  * Prior neoadjuvant or adjuvant therapy is allowed if the disease-free interval has been longer than 6 months
* No other concurrent chemotherapy
* No concurrent combination anti-retroviral therapy for HIV-positive patients
* No concurrent routine prophylaxis with filgrastim (G-CSF)
* No other concurrent antineoplastic agents, including chemotherapy, radiation therapy, or biologic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-08; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura W. Goff, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (5):
- United States (5):
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from August 2007 to March 2011.
Pre-assignment Details: Forty-two patients signed consent, 9 of which were found to be ineligible to participate in the study.
Groups:
- 5-FU, Leucovorin, Oxaliplatin: Patients who have TSER*2/*2 or TSER*2/*3 genotypes will receive the modified FOLFOX-6 treatment. Patients homozygous for TSER*3 will not be included in study.
  * FOLFOX-6 chemotherapy: oxaliplatin IV in 500 ml D5W over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 5 minutes and then continuously over 46 hours on days 1 and 15.
  * Treatment courses repeat every 2 weeks +/- 3 days (2 treatments per cycle) in the absence of unacceptable toxicity or disease progression. Disease assessments will be performed after 8 weeks (2 cycles) of treatment.
Period: Overall Study
Arm/Group | 5-FU, Leucovorin, Oxaliplatin
Started | 33 (two patients withdrew before treatment; one withdrew after treatment)
Completed | 5
Not Completed | 28
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Not completed — disease progression | 9
Not completed — other complicating disease | 2
Not completed — patient went to radiation treatment | 1
Not completed — patients moved to the "no tx" group | 6

BASELINE CHARACTERISTICS:
Groups:
- Oxaliplatin + Leucovorin + 5-Fluorouracil: Patients receive oxaliplatin IV over 2 hours, leucovorin calcium intravenously (IV) over 2 hours, and fluorouracil IV over 5 minutes and then continuously over 46 hours on days 1 and 15. Courses repeat every 2 weeks in the absence of unacceptable toxicity or disease progression.
Arm/Group | Oxaliplatin + Leucovorin + 5-Fluorouracil
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Each Response in "Good Risk" Genotype (Thymidylate Synthase Promoter Enhancer Region [TSER]*2/*2 or TSER*2/*3 Genotype [Low TS Expression])
Description: Per RECIST criteria v. 1.0: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, progressive disease (PD) > 20% increase in the sum of the LD of target lesions or appearance of new lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions. This is a one-time assessment.
Time Frame: every 8 weeks to progression
Population: Patients available for measurement of response. All patients who received Oxaliplatin + Leucovorin + 5-Fluorouracil are in the heterozygous "good risk" genotype group. One patient was not evaluable for response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin + Leucovorin + 5-Fluorouracil
Number analyzed (Participants) | 24
participants
  Complete Response | 0
  Partial Response | 9
  Progressive Disease | 1
  Stable Disease | 14

ADVERSE EVENTS:
Arm/Group | Oxaliplatin + Leucovorin + 5-Fluorouracil
Serious Adverse Events (participants affected / at risk) | 14/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin + Leucovorin + 5-Fluorouracil (N=24)
constipation (Gastrointestinal disorders) | 3 (6)
distension/bloating, abdominal (Gastrointestinal disorders) | 1 (2)
dysphagia (Gastrointestinal disorders) | 3 (6)
fever (in the absence of neutropenia, where neutropenia is defined as ANC < 1.0 x 10e9/L) (General disorders) | 1 (2)
nausea (Gastrointestinal disorders) | 4 (6)
obstruction, GU-ureter (Renal and urinary disorders) | 1 (2)
pain-abdomen NOS (Gastrointestinal disorders) | 6 (10)
urinary retention (Renal and urinary disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 3 (4)
INR (international normalized ratio of prothrombin) (Blood and lymphatic system disorders) | 1 (2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1)
death not associated with CTCAE-disease progression NOS (General disorders) | 2 (2)
infection with normal ANC or Grade 1 or 2 neutrophils-skin (cellulitis) (Skin and subcutaneous tissue disorders) | 1 (2)
supraventricular and nodal arrhythmia-atrial fibrillation (Cardiac disorders) | 2 (3)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin + Leucovorin + 5-Fluorouracil (N=24)
albumin, serum-low (Metabolism and nutrition disorders) | 17 (29)
alkaline phosphatase (Investigations) | 10 (13)
ALT/SGPT (serum glutamine pyruvic transminase) (Investigations) | 11 (15)
anorexia (Metabolism and nutrition disorders) | 8 (8)
ascites (non-malignant) (Gastrointestinal disorders) | 3 (4)
AST, SGOT (serum glutamine oxaloacetic transminase) (Investigations) | 11 (13)
bilirubin (hyperbilirubinemia) (Hepatobiliary disorders) | 2 (3)
calcium, serum-low-hypocalcemia (Metabolism and nutrition disorders) | 10 (14)
constipation (Gastrointestinal disorders) | 7 (11)
creatine (Investigations) | 2 (3)
dermatology/skin-other (Skin and subcutaneous tissue disorders) | 2 (3)
diarrhea (Gastrointestinal disorders) | 8 (14)
distension/bloating, abdominal (Gastrointestinal disorders) | 6 (6)
dizziness (Nervous system disorders) | 2 (2)
dysphagia (Gastrointestinal disorders) | 3 (3)
edema-limb (Musculoskeletal and connective tissue disorders) | 3 (3)
fatigue (General disorders) | 12 (17)
glucose, serum-high-hyperglycemia (Metabolism and nutrition disorders) | 11 (21)
heartburn/dyspepsia (Gastrointestinal disorders) | 2 (2)
hemoglobin (Investigations) | 22 (33)
insomnia (Psychiatric disorders) | 3 (4)
leukocytes (total WBC) (Blood and lymphatic system disorders) | 14 (32)
lymphopenia (Blood and lymphatic system disorders) | 9 (19)
metabolic/laboratory-other (Investigations) | 2 (2)
mood alteration-anxiety (Psychiatric disorders) | 2 (2)
mood alteration-depression (Psychiatric disorders) | 2 (2)
mucositis/stomatitis (clinical exam)-oral cavity (Gastrointestinal disorders) | 4 (6)
Mucositis/stomatitis (functional/symptomatic)-oral cavity (Gastrointestinal disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 15 (22)
neuropathy - sensory (Nervous system disorders) | 14 (39)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 12 (40)
pain-abdomen NOS (Gastrointestinal disorders) | 8 (16)
Pain-extremity-limb (Musculoskeletal and connective tissue disorders) | 2 (2)
pain-other (General disorders) | 2 (2)
platelets (Blood and lymphatic system disorders) | 14 (32)
potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6 (10)
rash-hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (2)
sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 (8)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 8 (8)
vision/blurred vision (Eye disorders) | 3 (3)
vomiting (Gastrointestinal disorders) | 7 (11)
weight loss (Investigations) | 2 (2)
fever in the absence of neutropenia, where neutropenia is defined as ANC < 1.0 x 12e9/L (Infections and infestations) | 2 (2)
infection with normal ANC or Grade 1 or 2 neutrophils-abdomen NOS (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes